CLINICAL TRIAL: NCT01093469
Title: An Investigator Blinded, Randomized, Controlled Study Comparing the Efficacy and Cost-Effectiveness of Aquaphor Healing Ointment, Atopiclair Nonsteroidal Cream (MAS063DP) and EpiCeram Skin Barrier Emulsion in Children With Mild to Moderate Atopic Dermatitis
Brief Title: Comparing Aquaphor to Atopiclair and EpiCeram in Children With Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00009130
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Wake Forest; Dermatology; Skin; Over-the-counter; Moisturizer; Children
MeSH Terms: conditions — Dermatitis, Atopic | interventions — MAS063DP; EpiCeram

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aquaphor Healing Ointment (Experimental): Aquaphor Healing Ointment three times daily to atopic dermatitis
  Interventions: Other: Aquaphor Healing Ointment
- Atopiclair Nonsteroidal Cream (Active Comparator): Atopiclair Nonsteroidal Cream three times daily to atopic dermatitis
  Interventions: Drug: Atopiclair Nonsteroidal Cream
- EpiCream Skin Barrier Emulsion (Active Comparator): EpiCream Skin Barrier Emulsion three times daily to atopic dermatitis
  Interventions: Drug: EpiCeram

INTERVENTIONS:
Drug: Atopiclair Nonsteroidal Cream
  Other Names: MAS063DP
  Arms: Atopiclair Nonsteroidal Cream
Other: Aquaphor Healing Ointment
  Arms: Aquaphor Healing Ointment
Drug: EpiCeram
  Other Names: BRC-Cer
  Arms: EpiCream Skin Barrier Emulsion

SUMMARY:
The purpose of this study is to compare the efficacy and cost effectiveness of Aquaphor Healing Ointment, Atopiclair and EpiCeram as a monotherapy in mild to moderate AD.

The investigators hypothesize that no statistical difference will exist in the efficacy between an over-the-counter moisturizer, Aquaphor Healing Ointment, compared to prescription devices Atopiclair and EpiCeram in treating mild to moderate AD. Therefore, Aquaphor will be most cost-effective than Atopiclair or EpiCeram.

DETAILED DESCRIPTION:
The primary objective is to compare the efficacy of Aquaphor Healing Ointment, Atopiclair Nonsteroidal Cream and EpiCeram Skin Barrier Emulsion in children with mild to moderate atopic dermatitis. The secondary objective is to compare the cost-effectiveness of these products. A significant difference exists in the cost of these products; therefore, if our hypothesis is proved correct - that Aquaphor will be just as efficacious as the more expensive counterparts Atopiclair and EpiCeram - this could have a significant impact on the overall cost of treating atopic dermatitis.

This is a single center, investigator blinded, randomized, prospective controlled study of subjects with mild to moderate atopic dermatitis. The study is intended to compare the efficacy of Aquaphor Healing Ointment, Atopiclair Nonsteroidal Cream and the EpiCeram Skin Barrier Emulsion used three times a day in treating mild to moderate atopic dermatitis. All subjects will receive active study medication and will return to study center for efficacy and safety assessments at Days 7 and 21. Approximately 50 subjects will be enrolled in order to obtain 39 completed subjects that will be randomized 1:1:1 (13 to receive Aquaphor, 13 to receive Atopiclair and 13 to receive EpiCeram) according to standard randomization tables. Efficacy will be measured through Investigator's Global Assessment, BSA involvement, Investigator Global Assessment of Improvement, Eczema Area and Severity Index and 100-pt Visual Analog Score for pruritis. Subjects will complete a Subject Global Assessment of Improvement and a drug diary to monitor for compliance. Cost benefit analysis will be calculated as cost in dollars for change in outcome according to EASI, BSA and VAS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with mild to moderate atopic dermatitis, 2-17 years of age, that agree to participate and provide written consent (and assent if applicable)
* Have an investigator Global Assessment of mild to moderate atopic dermatitis (IGA rating of 2-3 in the Investigator Global Assessment)
* Percentage of overall body surface area of involvement (BSA) must be > 1% and may include facial and intertriginous skin.

Exclusion Criteria:

* Use within 4 weeks of baseline of systemic anti-inflammatory medication, which may influence study outcome, such as systemic corticosteroids.
* Application or use within 2 weeks of baseline of topical corticosteroid medications or topical anti-inflammatory medication, which may influence study outcome.
* Presence of a concurrent medical condition, which is determined by the investigator to potentially interfere with study outcomes or patient assessments.
* Introduction of any other prescription medication, topical or systemic, for atopic dermatitis while participating int he study (oral antihistamines will be allowed, so long as they are neither initiated nor discontinued during the course of this study)
* Amount of disease involvement that would require >60gm of cream in a 1 week period
* Subjects with known allergy or sensitivity to Aquaphor Healing Ointment, Atopiclair or EpiCeram or components therein.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Fleischer, MD, Principal Investigator — Wake Forest University Health Sciences Department of Dermatology
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller DW, Koch SB, Yentzer BA, Clark AR, O'Neill JR, Fountain J, Weber TM, Fleischer AB Jr. An over-the-counter moisturizer is as clinically effective as, and more cost-effective than, prescription barrier creams in the treatment of children with mild-to-moderate atopic dermatitis: a randomized, controlled trial. J Drugs Dermatol. 2011 May;10(5):531-7. PMID 21533301

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aquaphor Healing Ointment | Atopiclair Nonsteroidal Cream | EpiCream Skin Barrier Emulsion
Started | 13 | 13 | 13
Completed | 13 | 13 | 12
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aquaphor Healing Ointment | Atopiclair Nonsteroidal Cream | EpiCream Skin Barrier Emulsion | Total
Number analyzed (Participants) | 13 | 13 | 13 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 13 | 13 | 39
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 22
  Male | 6 | 6 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 11 | 13 | 12 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 6 | 7 | 14
  White | 10 | 7 | 6 | 23
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 13 | 39

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment of Improvement
Description: This measures the overall response to treatment and quantifies disease on a 6 point scale from "completely clear" to "worsening of disease".0= Completely clear: except for possible residual hyperpigmentation, 1= Almost clear: very significant clearance (about 90%), 2 = Marked improvement: significant improvement (about 75%), 3= Moderate improvement: intermediate between slight and marked; representing about 50% improvements , 4= Slight improvement: some improvement (about 25%); however, significant disease remaining, 5 = No change from baseline, 6 = Worse
Time Frame: Day 21
Measure: Median (Standard Error); unit: units on a scale
Arm/Group | Aquaphor Healing Ointment | Atopiclair Nonsteroidal Cream | EpiCream Skin Barrier Emulsion
Number analyzed (Participants) | 13 | 13 | 12
units on a scale | 2 (1.7) | 2 (2.0) | 2 (1.9)

ADVERSE EVENTS:
Arm/Group | Aquaphor Healing Ointment | Atopiclair Nonsteroidal Cream | EpiCream Skin Barrier Emulsion
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 2/13 | 2/13 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aquaphor Healing Ointment (N=13) | Atopiclair Nonsteroidal Cream (N=13) | EpiCream Skin Barrier Emulsion (N=13)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
MRSA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Worsening ATD (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less